CLINICAL TRIAL: NCT00803400
Title: Efficacy of Aerobic Exercise Added to Alprazolam in Panic Disorder Treatment: a Clinical Randomized Trial
Brief Title: Efficacy of Aerobic Exercise Added to Alprazolam in Panic Disorder Treatment
Acronym: AEIPDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr.Marcelo Rudelir, Ph D, University of Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDHFMEDUBA0709
Record Dates: First submitted 2008-11-07; First posted 2008-12-05 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Panic Disorder
Keywords: Panic disorder; Exercise; Alprazolam; Aerobic
MeSH Terms: conditions — Panic Disorder; Motor Activity | interventions — Alprazolam; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alprazolam (Active Comparator): Patients assigned to the pharmacological plan
  Interventions: Drug: Alprazolam
- Alprazolam + Aerobic exercise (Active Comparator): Patients assigned to mix plan
  Interventions: Drug: Alprazolam + Aerobic exercise

INTERVENTIONS:
Drug: Alprazolam — The patients assigned to the pharmacological plan will receive 4 mg alprazolam daily for 12 weeks. Two weeks after the first interview they have their first baseline psychiatric control, where all the patients are tested.
  Then, at the same visit, all the patients are indicated 4 mg of alprazolam. The dose is gradually increased from 1 to 4 mg along the first week of treatment. The test is repeated during weeks 2, 4, 8 and 12.
  Other Names: Non exercise group
  Arms: Alprazolam
Drug: Alprazolam + Aerobic exercise — The patients assigned to exercise have to pass an ergometric test to determine their functional capacity expressed in METs for future exercise indication.
  Two weeks after the first interview they have their first baseline psychiatric control and at the same time they are indicated a 4 mg dose of alprazolam, gradually increased from 1 to 4 mg along the first week of treatment. The test is repeated during weeks 2, 4, 8 and 12.
  Then they follow a protocolized aerobic exercise plan for this study during 12 weeks.
  The type of selected exercise consists of a rapid walk for 30 minutes divided in stages.
  After each stage the patient has to control his own heart frequency that has to be between 50 and 75% of their maximum to assure an aerobic condition (American Cardiological Association).
  Other Names: Exercise group
  Arms: Alprazolam + Aerobic exercise

SUMMARY:
The purpose of this study is to determine whether the combination of aerobic physical exercise and alprazolam in patients with panic disorder has a better therapeutic response than the treatment with alprazolam alone.

DETAILED DESCRIPTION:
We have observed in our clinical practice that patients who practiced aerobic physical exercise had faster remissions and better improvement in their treatments that those who did not. There are also some scientific studies that included physical exercise in the treatment for panic disorder and compared them to other single pharmacological treatments.

So our objective will be to compare the efficacy of a pharmacological monotherapy (alprazolam), that is one of the options for the pharmacological treatment of panic disorder, with other treatment such as the combination of aerobic physical exercise and alprazolam, and to determine if this combination results in a better therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with panic disorder scored between 20 and 30 by the Hamilton Anxiety Rating Scale/14. (Baseline scale scores were measured during the first interview and diagnoses were made by a psychiatrist using the Structured Clinical Interview for DSM IV).
* Good physical health and normal results determined on a previous physical examination and routine laboratory tests (renal, hepatic, hematological and thyroid function).
* Patients who completed a written informed consent form (which was obtained from every included patient and had been fully explained before the procedure).

Exclusion Criteria:

* A history of some kind of recent somatic disease.
* Diagnosis of some other type of associated or psychiatric disease of axis I of DSM IV, such as affective disorders, drug dependency.
* Hamilton Anxiety Scale lower than 20 points or higher than 30.
* Use of some other type of medication or treatment (including psychotherapy) or having received it during last past 3 months.
* Patients who could not complete the clinical examination
* Patients who have not accepted to complete or sign the written informed consent.
* Pregnant patients or in lactation. (A pregnancy test was performed for women in fertile age)
* Patients with history of rejection to the used drug.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo G Rudelir, MD, Principal Investigator — Psychiatry and Mental Health Department at University of Buenos Aires
Locations (1):
- Psychiatry Academic Unit at J.A.Fernandez Hospital, University of Buenos Aires Medicine School Department of Mental Health, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toro Martinez E, Rudelir M. [Assessment of suicide risk: clinical and legal aspects]. Vertex. 2005 May-Jun;16(61):196-205. Spanish. PMID 15957014
- See also: Psychiatry and Mental Health Department at University of Buenos Aires — https://www.fmed.uba.ar/index.php/departamentos_y_catedras/departamento-de-psiquiatria-y-salud-mental/autoridades-y-cuerpo-docente

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 180 patients were preselected for the study and 150 were eligible for the study. They were outpatients from the office practice and were recruited from March 2005 to July 2007.
Pre-assignment Details: 30 selected patients were not included: 12 did not match the 20 points for the Hamilton Anxiety Scale; 10 had history of medical diseases (5 of hypothyroidism, 4 of hypertension, and 1 of chronic fatigue syndrome); 8 had other associated psychiatric diseases: (5 had major depressive disorder and 3 had social anxiety disorder).
Groups:
- Alprazolam: Pacients receiving only alprazolam
- Alprazolam + Aerobic Exercise: Pacients receiving alprazolam + aerobic exercise
Period: Overall Study
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise
Started | 75 | 75
Completed | 55 | 51
Not Completed | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Alprazolam: Patients receiving only alprazolam
- Alprazolam + Aerobic Exercise: Patients receiving alprazolam + aerobic exercise
- Total: Total of all reporting groups
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.01 (8.07) | 35.68 (7.67) | 34.85 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  Argentina | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Participants´Endpoint Change From Baseline in Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale is a test that consists of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe).
  Each of the 14 items measure both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety)with a total score range of 0-56, where 17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise
Number analyzed (Participants) | 75 | 75
Units on a scale | 22.59 (2.09) | 22.73 (1.98)
Statistical Analysis 1: Comparison: Alprazolam vs Alprazolam + Aerobic Exercise; A p-value less than 0.05 (≤ 0.05) is statistically significant. It indicates strong evidence against the null hypothesis, as there is less than a 5% probability the null is correct (and the results are random); Test type: Other; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 1

2. Secondary Outcome: Participants´Endpoint Change From Baseline in Clinical Global Impression Severity Scale (CGI-S)
Description: The Clinical Global Impression Severity scale is a 7 point ordinal scale that rates the severity of the patient's illness, assessing on the severity of a patient's mental illness. It ranges from 1 to 7 (1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; 7, extremely ill).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Alprazolam: Patients only receiving alprazolam
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise
Number analyzed (Participants) | 75 | 75
Units on a scale | 4.05 (0.23) | 4.06 (0.24)

3. Secondary Outcome: Participants´Endpoint Change From Baseline in Clinical Global Impression Improvement Scale (CGI-I)
Description: The Clinical Global Impression Improvement Scale is a 7 point ordinal scale that assesses how much the patient's illness has improved or worsened relative to a baseline state before the intervention. Rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Baseline and 12 weeks
Population: Patients with history of Panic Disorder
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise
Number analyzed (Participants) | 55 | 51
Score on a scale | 2.70 (0.62) | 1.86 (0.60)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 weeks
Description: Definition of adverse events are similar of those taken from clinicaltrials.gov
Arm/Group | Alprazolam | Alprazolam + Aerobic Exercise
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 32/75 | 39/75
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alprazolam (N=75) | Alprazolam + Aerobic Exercise (N=75)
Somnolence (Nervous system disorders) | 28 (52) | 34 (60)
Dizziness (Nervous system disorders) | 4 (8) | 5 (9)

LIMITATIONS AND CAVEATS:
Panic patients may sometimes be reluctant to use medication. This could lead to early drop outs.

Possible difficulties in following the exercise protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes